CLINICAL TRIAL: NCT01604044
Title: Highly Purified Menotropin (HP-hMG) Versus Recombinant FSH (rFSH) Plus Recombinant LH (rLH) in Intrauterine Insemination Cycles in Women ≥35 Years: a Prospective Randomized Trial.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Rosanna Apa, professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Meropur2009
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female

ARMS (2):
- HP-hMG (Active Comparator)
  Interventions: Drug: Meropur 150 a day
- rFSH plus rLH (Active Comparator)
  Interventions: Drug: Gonal-f 150 plus Luveris 150

INTERVENTIONS:
Drug: Meropur 150 a day — one subcutaneous injection a day
  Arms: HP-hMG
Drug: Gonal-f 150 plus Luveris 150 — one subcutaneous injection a day
  Arms: rFSH plus rLH

SUMMARY:
This study evaluates the effects of different therapies in ovulation induction in Intrauterine Insemination Cycles.

ELIGIBILITY:
Inclusion Criteria:

* women with story of infertility sine causa and mild-moderate male factor
* regular ovulatory menstrual cycles
* BMI ≤27 kg/m2
* normal day 3 hormonal pattern
* bilateral tubal patency

Exclusion Criteria:

* mono/bilateral tubal occlusion,
* severe male factor
* polycystic ovarian syndrome or any systemic disease or endocrine or metabolic abnormalities
* pelvic inflammatory disease
* endometriosis
* sexual organ malformations
* neoplasms or breast pathology incompatible with gonadotropin stimulation.

Ages: 35 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 579 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy rate | 12 weeks

SECONDARY OUTCOMES:
number of cancelled cycles for low or no response, the number of interrupted cycles for high risk of OHSS and multiple pregnancies | 30 days

OTHER OUTCOMES:
duration of stimulation, total gonadotropin dose, number of midsize follicles, dominant follicles, E2 levels, endometrial thickness on hCG day, Progesterone levels, endometrial thickness on the midluteal phase. | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Agostino Gemelli, Rome, Rome, Italy

REFERENCES:
- [Derived] Moro F, Scarinci E, Palla C, Romani F, Familiari A, Tropea A, Leoncini E, Lanzone A, Apa R. Highly purified hMG versus recombinant FSH plus recombinant LH in intrauterine insemination cycles in women >/=35 years: a RCT. Hum Reprod. 2015 Jan;30(1):179-85. doi: 10.1093/humrep/deu302. Epub 2014 Nov 14. PMID 25398971